CLINICAL TRIAL: NCT02064725
Title: A Phase II Study of Sodium Cridanimod in Conjunction With Progestin Therapy in Patients With Progesterone Receptor Negative Recurrent or Persistent Endometrial Carcinoma
Brief Title: Virexxa (Sodium Cridanimod) w/Progestin Therapy in Pts w/Progesterone Receptor Neg Recurrent/Persistent Endometrial CA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kevelt AS (Industry)
Collaborators: Pharmasyntez (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX-EC-2-2013
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent or Persistent Endometrial Carcinoma
Keywords: Endometrial cancer; Recurrent or persistent endometrial carcinoma; Progesterone Receptor Negative; Sodium cridanimod; Virexxa
MeSH Terms: conditions — Recurrence; Endometrial Neoplasms | interventions — 10-carboxymethyl-9-acridanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium cridanimod (Experimental): Sodium cridanimod in combination with megestrol acetate or medroxyprogesterone acetate. Treatment period is 12 months; patients will be followed for another 12 month period or to disease progression whichever occurs first.
  Interventions: Drug: Sodium cridanimod

INTERVENTIONS:
Drug: Sodium cridanimod — Eligible patients will be enrolled into the study and administered sodium cridanimod (500 mg i.m./ twice a week) in combination with megestrol acetate (160 mg p.o./ day) or medroxyprogesterone acetate (200 mg p.o./ day).
  Other Names: Virexxa

SUMMARY:
This is an open label, multi-center, single arm phase II study. The study will investigate the efficacy of sodium cridanimod in conjunction with progestin therapy in a population of patients with recurrent or persistent PrR-negative endometrial cancer.

DETAILED DESCRIPTION:
This is an open label, multi-center, single arm phase II study. The study will investigate the efficacy of sodium cridanimod in conjunction with progestin therapy in a population of patients with recurrent or persistent PrR-negative endometrial cancer.

Eligible patients will be enrolled into the study and administered sodium cridanimod in combination progestin therapy. Objective responses will be assessed at 12 week intervals. Patients will be treated for a 12 month period, followed by an additional 12 month follow up period or to disease progression whichever occurs first.

Important objectives of the study are to investigate the effect of sodium cridanimod in conjunction with progestin therapy on the level of PrR in tumor tissue and how this correlates to efficacy. To accomplish this objective, some of the patients enrolled in the study will undergo two tumor biopsies that will allow measurement of PrR levels in the tumor tissue before the treatment and after 4 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients age 18 and older;
* Histologically confirmed papillary serous adenocarcinoma or endometrioid type of endometrial carcinoma (histological documentation of recurrence is not required);
* Patient has documented evidence of PrR negative endometrial cancer. PrR negativity can be determined by immunohistochemistry. The tumor is considered PrR negative if the number of PrR positive cells is less than 1% determined by immunohistochemistry;
* Availability of tumor tissue sample that can be used for assessment of PrR levels with the use of immunohistochemistry;
* Recurrent or persistent (after the failure of chemotherapy) disease that cannot be treated with surgery or radiotherapy;
* Documented disease progression after a platinum based chemotherapy in patients for whom administration of taxanes and anthracyclines is not planned. Progression must fulfill one of the following criteria:

  * Progression has occurred within 30 days of platinum based chemotherapy consisting of minimum of two cycles of cisplatin-based (≥60 mg/m2/cycle) or carboplatin-based (≥300 mg/m2/cycle, or area under the time-concentration curve ≥4) chemotherapy.
  * Progression after neoadjuvant or adjuvant platinum based chemotherapy if the recurrence occurred while on neoadjuvant/adjuvant chemotherapy or within 6 months since the last administration of such therapy.
* Measurable disease as defined by RECIST 1.1 criteria;
* At least one "target lesion" to be used to assess response, as defined by RECIST 1.1 criteria;
* Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented;
* GOG performance status 0-2;
* Glomerular filtration rate ≥ 50 mL/min;
* Total bilirubin normal;
* AST ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN for patients with liver metastases);
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases);
* Albumin ≥ 3.0 mg/dL;
* Ability to take oral medication;
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Evidence of histology of the tumor other than papillary serous adenocarcinoma or endometrioid type of endometrial carcinoma or mixed histology of the tumor;
* History of hormonal therapy for endometrial carcinoma for more than 3 months;
* History of use of progestins for a period of longer than 3 months for any indication, including endometriosis;
* Concurrent maintenance corticosteroids;
* Concurrent oral contraceptives/ Fertile patients must use effective barrier contraception;
* Pregnancy as determined by pregnancy test or nursing;
* History of bleeding (i.e. disseminated intravascular coagulation or clotting factor deficiency);
* Prior major surgery less than 4 weeks prior to the start of the study;
* Concurrent serious illness which, in the opinion of the investigator, would place the patient at unreasonable risk from study therapy;
* Previous malignancy less than 3 years ago other than in situ carcinoma of the cervix, basal cell carcinoma or squamous carcinoma of the skin;
* History of allergic reactions or idiosyncrasy attributed to progestins or compounds of similar chemical structure to sodium cridanimod or lidocaine;
* Known brain metastases;
* Other concurrent investigational agents;
* Other concurrent anticancer therapies.
* Known carrier of HIV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 months

SECONDARY OUTCOMES:
Progression-free survival | 24 months
Time to response | 12 months
Time to progression | 24 months
Overall survival | 24 months
Overall Disease Control Rate | 24 months

OTHER OUTCOMES:
Progesterone receptor (PrR) levels | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura L. Douglass, Study Director — Kevelt AS
Locations (21):
- United States (4):
  - Physicians Research Group, San Jose, California
  - St. Jude Hospital Yorba Linda, St. Joseph's Heritage Healthcare, Santa Rosa, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
- Belarus (4):
  - Brest Regional Clinical Hospital, Brest
  - Minsk City Clinical Oncology Dispensary, Minsk
  - N.N. Alexandrov National Cancer Centre of Belarus, Minsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Oncology, Olomouc
- Slovakia (3):
  - Oncology Institute of Saint Alzbeta, Bratislava
  - Poko Poprad, s.r.o., Poprad
  - University Hospital Trencin, Trenčín
- Ukraine (7):
  - Cherkasy Regional Oncology Dispensary, Cherkasy
  - Municipal Institution of Dnipropetrovsk Regional Rada, Dnipropetrovsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - S.P. Grigoryeva Institute of Medical Radiology, Kharkiv
  - Kherson Regional Oncological Dispensary, Kherson
  - Sumy State University, Sumy
  - Vinnitsa Regional Clinical Oncology Center, Vinnitsa